CLINICAL TRIAL: NCT01296607
Title: Effects of Urocortins on Forearm Arterial Blood Flow in Healthy Volunteers
Brief Title: Effects of Urocortins on Forearm Arterial Blood Flow in Healthy Volunteers - Protocol 4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SV.Protocol 4
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Disease; Heart Failure
Keywords: Pharmacodynamics; Pharmacokinetics; Urocortin 2; Urocortin 3; Reproducibility; Onset/ Offset; Forearm blood flow; Plethysmography; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure | interventions — Urocortins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urocortin 2 (Other): This arm studies the onset/ offset of action and the reproducibility of effect on forearm blood flow of of intra-arterial Urocortin 2 in the presence and absence of a saline washout between incremental doses.
  Interventions: Drug: Urocortin 2
- Urocortin 3 (Other): This arm studies the onset/ offset of action and the reproducibility of effect on forearm blood flow of of intra-arterial Urocortin 3 in the presence and absence of a saline washout between incremental doses.
  Interventions: Drug: Urocortin 3

INTERVENTIONS:
Drug: Urocortin 2 — Protocol 4a: Onset/Offset protocol: (Visits 1 or 3)
  Following a 20-minute period of saline infusion for equilibration of the set-up, subjects will receive incremental doses of Urocortin 2 in the presence of a saline washout between each dose.
  Urocortin 2 will be infused at 3.6, 12, 36 and 120 pmol/min (15, 50, 150 and 498 nanograms/min) to achieve estimated end-organ concentrations of 0.6, 2, 6 and 20 micrograms/L respectively.
  Protocol 4b: Reproducibility protocol (Visit 2 or 4)
  Following a 20-minute period of saline infusion for equilibration of the set-up, subjects will receive ascending doses of urocortin 2 in the absence of saline washout between each dose. This protocol aims to assess the reproducibility of the vasodilatory effect of urocortin 2 on repeated dosing. The doses used for this protocol will be identical to Protocol a.
  Arms: Urocortin 2
Drug: Urocortin 3 — Protocol 4a: Onset/ Offset protocol: (Visit 1 or 3)
  Following a 20-minute period of saline infusion for equilibration of the set-up, subjects will receive incremental doses of Urocortin 2 or Urocortin 3 in the presence of a saline washout between each dose.
  Urocortin 3 will be infused at 1200, 3600, 12000 and 36000 pmol/min (5, 15, 50 and 150 micrograms/min) to achieve estimated end organ concentrations of 199, 600, 2000 and 6000 micrograms/L respectively.
  Protocol 4b: Reproducibility protocol (Visit 2 or 4)
  Following a 20-minute period of saline infusion for equilibration of the set-up, subjects will receive ascending doses of urocortin 3 in the absence of saline washout between each dose. This protocol aims to assess the reproducibility of the vasodilatory effect of 3 on repeated dosing. The doses used for this protocol will be identical to Protocol a.
  Arms: Urocortin 3

SUMMARY:
Impairment of the heart's pumping capacity (heart failure) remains a major clinical problem with a poor prognosis and the search for novel treatments remains an important area of research.

Urocortins are proteins that appear to increase blood flow and heart pumping activity. There has been particular interest in the role of Urocortins 2 & 3 (subtypes of Urocortins) in heart failure.

In this study, we will examine the pharmacokinetics and pharmacodynamics (in particular the onset-offset of action and reproducibility of vasodilator effects) of Urocortins 2 & 3 on forearm arterial blood flow healthy volunteers.

Utilising the well-established technique of 'forearm venous occlusion plethysmography', we will be able to focus on the local effects of urocortins on arterial blood flow in forearm vessels, without affecting this system in the body as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 - 65 years (inclusive)

Exclusion Criteria:

* Lack of informed consent- Age <18 years > 65 years
* Current involvement in a clinical trial
* Severe or significant co-morbidity including bleeding diathesis, renal or hepatic failure
* Smoker
* History of anaemia
* Recent infective/inflammatory condition
* Recent blood donation (prior 3 months)
* Positive baseline urine test for drugs of abuse (including cannabinoids, benzodiazepines, opiates, cocaine and amphetamines)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow | 3.5 hours
  Difference in forearm blood flow in response to increasing doses of Urocortin 2 and Urocortin 3 in the presence and absence of saline washout between doses

SECONDARY OUTCOMES:
Plasma Urocortin 2 and 3 levels | 3.5 hours
  Change in plasma levels of Urocortin 2 and 3 in response to intra-arterial infusion of Urocortin 2 and 3 respectively.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD, FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Wellcome Trust Clinical Research Facility, Royal Infirmary of Edinburgh, Edinburgh, Mid Lothian, United Kingdom

REFERENCES:
- [Derived] Venkatasubramanian S, Griffiths ME, McLean SG, Miller MR, Luo R, Lang NN, Newby DE. Vascular effects of urocortins 2 and 3 in healthy volunteers. J Am Heart Assoc. 2013 Jan 31;2(1):e004267. doi: 10.1161/JAHA.112.004267. PMID 23525432